CLINICAL TRIAL: NCT05422547
Title: Role of Immunoscore® in Stage II-III Colorectal Cancer
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: D'Or Institute for Research and Education (Other)
Collaborators: HalioDx (Industry); Diagnosticos da America SA (Unknown)
Responsible Party: Sponsor
Other Study IDs: Immunoscore®
Record Dates: First submitted 2022-05-30; First posted 2022-06-16 (Actual); Last update posted 2022-06-16 (Actual); Status verified 2022-06

CONDITIONS: Colon Adenocarcinoma
Keywords: colorectal cancer; colon carcinoma; immunoscore; immune response; predictive markers; prognostic markers; tumour microenvironment
MeSH Terms: conditions — Colonic Neoplasms; Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Colorectal cancer resection surgical biospecimen
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Immunoscore Colon Test — Immunoscore® is a tissue-based immune test that measures the host's immune response at the site of the tumor. It is performed on formalin-fixed paraffin-embedded (FFPE) tumor tissue samples from resections of localized colon cancer. The test uses whole slide imaging and artificial intelligence algorithms for assessment of the type, density, and location of T cells in FFPE tumor sections to determine an individual Immunoscore® for each patient.

SUMMARY:
The proposed study is a bidirectional analytical study, composed of a retrospective and a prospective cohorts. Patients with stage II - III colorectal cancer undergoing oncological surgery will be analyzed. The study will include a convenience sample of 100 individuals. Fifty cases will be included retrospectively and fifty prospectively.

The study aims to evaluate the benefit of using the Immunoscore test as a predictor of recurrence in patients with operated stage II-III colon tumors. It will also be evaluated the impact on oncologic decision and costs.

ELIGIBILITY:
Inclusion Criteria:

1. Anatomopathological diagnosis of colorectal adenocarcinoma
2. Stage II - III (AJCC 8th edition)
3. Patient undergoing surgery with curative intent

Exclusion Criteria:

1. Current or previous diagnosis (within the last 5 years) of another invasive primary malignant neoplasm, with the exception of non-melanoma skin neoplasm
2. Presence of distant metastatic disease evidenced in imaging tests

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Patients with stage II - III colorectal cancer undergoing oncological surgery.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2022-04-01 (Actual); Primary Completion 2022-12-30 (Estimated); Study Completion 2023-12-30 (Estimated)

PRIMARY OUTCOMES:
Tumour recurrence | 2 years
  Impact of Immunoscore stratification on tumor recurrence at 2 years

SECONDARY OUTCOMES:
Disease-free survival (DFS) | 5 years
  Impact of Immunoscore stratification on DFS at 5 years
Overall survival (OS) | 5 years
  Impact of Immunoscore stratification on OS at 5 years
DFS acoording tumor side | 3 years
  Impact of Immunoscore stratification on DFS in right and left tumors at 3 years
OS acoording tumor side | 3 years
  Impact of Immunoscore stratification on OS in right and left tumors at 3 years
Indication of adjuvant therapy | 6 months
  Percentage of patients who had an indication for adjuvant therapy through the evaluation of medical prescriptions
Biomarker measurements | 6 months
  Correlation of Immunoscore stratification with the KRAS, NRAS and BRAF status
Possible economic impact | 5 years
  Difference in monetary value due to Immuno Score stratification and chemotherapy indication

CONTACTS AND LOCATIONS:
Overall Officials: Paulo M Hoff, PhD, Study Chair — Instituto D'Or de Pesquisa e Ensino; Fernando A Soares, PhD, Study Chair — Instituto D'Or de Pesquisa e Ensino
Locations (2):
- Brazil (2):
  - Instituto D'Or de Pesquisa e Ensino - Brasília, Brasília, Federal District
  - Instituto D'Or de Pesquisa e Ensino - Rio de Janeiro, Rio de Janeiro

IPD SHARING:
Plan to Share IPD: No